CLINICAL TRIAL: NCT05664633
Title: A Randomized Clinical Trial to Determine the Effect of Transient Postoperative Urinary Retention Using Sugammadex (4 Mg X Kg) Versus Glycopyrrolate and Neostigmine (0.01 Mg/kg - 50mg/kg) in Patients Undergoing Vaginal Hysterectomies with and Without Pelvic Organ Prolapse Procedures: a Pilot Study
Brief Title: The Role of Sugammadex in Posotoperative Urinary Retention in Patients Undergoing Pelvic Floor Reconstructive Procedures
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: technical aspects - unable to continue with the study. Investigator left institution. No patients enrolled.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Omar Duenas Garcia, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2107367192
Record Dates: First submitted 2022-12-15; First posted 2022-12-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Urinary Retention
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Active Comparator): Sugammadex dose=4 mg x kg
  Interventions: Drug: Sugammadex
- Standard of Care (No Intervention): Standard of care= glycopyrrolate and neostigmine (0.01 mg/kg - 50mg/kg)

INTERVENTIONS:
Drug: Sugammadex — Sugammadex or G/N will be given at the end of the procedure once the surgeon communicates with the anesthesiologist. The surgeon will typically do this at the time of putting the closing sutures.
  Arms: Sugammadex

SUMMARY:
The Investigator will perform a single-institution randomized double-blinded controlled trial comparing intraoperative Sugammadex vs. standard dose of glycopyrrolate/neostigmine combination for participants undergoing a total vaginal hysterectomy with or without pelvic organ prolapse procedures under general endotracheal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* female patients undergoing a vaginal hysterectomy with the indications of pelvic organ prolapse or abnormal uterine bleeding

Exclusion Criteria:

* Patients who are already known to have voiding dysfunction
* Patients who have a contraindication or intolerance to any of the drugs used in the study
* Has a medical condition or surgical procedure that precludes reversal of neuromuscular block at the end of surgery.
* Has a neuromuscular disorder(s) that may affect neuromuscular block and/or trial assessments.
* Is dialysis-dependent or has severe renal insufficiency, defined as estimated creatinine clearance of <30 mL/min.
* Has or is suspected of having a personal history or family history (parents, grandparents, or siblings) of malignant hyperthermia.
* Has or is suspected of having an allergy (e.g., hypersensitivity and/or anaphylactic reaction) to study treatments or its/their excipients, to opioids/opiates, muscle relaxants or their excipients, or other medication(s) used during general anesthesia.
* Has received or is planned to receive toremifene within 24 hours before or within 24 hours after study medication administration.
* Has any condition that would contraindicate the administration of study medication.
* Is pregnant, is attempting to become pregnant, or is lactating.
* Is currently participating in or has participated in an interventional clinical trial (including any other current or ongoing trial with a sugammadex treatment arm) with an investigational compound or device within 30 days of signing the informed consent form of this current trial.
* Male patients
* Patients undergoing a conventional laparoscopic or robotic approach
* Patients having a midurethral sling in addition to the vaginal hysterectomy
* Patients declining to participate in the study
* Patients allergic to any of the drugs used in the study (sugammadex, neostigmine and/or glycopyrrolate)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Void Test (Pass) | Up to 4 hours postop
  Number of patients that Pass the Void Test. Once the patients are oriented and before leaving PACU, their bladder will be backfilled with 300 ccs of normal saline or at capacity. Then 30 minutes will be given to void. The voided volume will be measured using a toilet hat, and the post-void residual will then be measured using a bladder scanner.
Void Test (Fail) | Up to 4 hours post-op
  Number of patients that Fail the Void Test. Once the patients are oriented and before leaving PACU, their bladder will be backfilled with 300 ccs of normal saline or at capacity. Then 30 minutes will be given to void. If the patients are unable to void or if the post-void residual is > than 100 ml by bladder scanner, then it will be considered that those patients failed the voiding trial

CONTACTS AND LOCATIONS:
Overall Officials: Omar Duenas Garcia, MD, Principal Investigator — WVU

IPD SHARING:
Plan to Share IPD: No